CLINICAL TRIAL: NCT06920355
Title: Community Pharmacy Produce Prescriptions (CP3): Design, Implementation, and Evaluation of a Produce Prescription Program in Community Pharmacies
Brief Title: Community Pharmacy Produce Prescriptions
Acronym: CP3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Association of Chain Drug Stores (Industry)
Responsible Party: Principal Investigator, Dariush Mozaffarian, Director, Food is Medicine Institute, Tufts University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00005176
Record Dates: First submitted 2025-02-26; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus Type 2; Hypertension
Keywords: Food is Medicine; Produce Prescriptions; Produce Rx; Community Pharmacy; Nutrition Security; Food Security; Nutrition Intervention; Food as Medicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Produce Prescription Group (Experimental)
  Interventions: Other: Produce Prescription; Behavioral: Nutrition Education

INTERVENTIONS:
Other: Produce Prescription — Each month, participants will receive a fixed amount of funds on the PRx card. Participants will be able to use these funds to purchase fruits, vegetables, beans, nuts, nut butters, seeds, plant-based oils, seafood, and yogurts from participating grocery stores. These funds will be provided through an electronic PRx benefit card that is activated after the initial baseline in-person visit is completed. The card will be reloaded monthly for a period of 6 months.
  Other Names: Produce Rx
Behavioral: Nutrition Education — Participating pharmacies/grocery chains will have Registered Dietitians (RD/RDN) on staff who can provide participants with nutrition education programs, coaching, and/or nudges.

SUMMARY:
The goal of this clinical trial is to generate evidence on the feasibility and effectiveness of community pharmacies as the implementers of a produce prescription program for adults with diabetes and/or hypertension. The main question this study plans to answer is if using community pharmacies as a point-of-service for improving nutrition and health is feasible and effective. The trial also explores the impact of the program on food security, nutrition security, diet quality and health and patient centered outcomes.

Participants will be enrolled in a produce prescription program to purchase healthy foods at the grocery store where they are currently receiving their pharmacy services. Participants will be asked to attend pharmacy visits to collect biometrics at two different time points and complete electronic surveys at three different time points.

DETAILED DESCRIPTION:
Produce prescription programs are an increasingly common Food is Medicine (FIM) intervention, with over 100 programs launched in US healthcare systems over the past decade. Mounting evidence from these programs suggests health-related benefits, including reductions in household food insecurity, increased consumption of fruits and vegetables, and improvements in clinical outcomes such as diastolic blood pressure, hemoglobin A1c, and body mass index.

Pharmacies routinely engage in vital screening and referral services, including monitoring blood glucose, blood pressure, cholesterol levels, and administering vaccinations, among other patient care services. However, the community pharmacy setting has remained a largely underutilized and understudied platform for advancing FIM. Historically, FIM interventions have been designed and delivered through hospitals, medical clinics, or community non-profit organizations. The next phase of FIM efforts involves expanding screening and referral for such programs to community pharmacies, including those affiliated or co-located with grocery stores. Community Pharmacy Produce Prescriptions study intervention will be delivered via a Produce Prescription (PRx) electronic benefit card. Each month, participants will receive a fixed amount of funds on the PRx card to purchase fruits, vegetables, beans, nuts, nut butters, seeds, plant-based oils, seafood, and yogurts from participating grocery stores. These funds will be provided after the initial baseline in-person visit is completed. The card will be reloaded monthly for a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Age 18 years or older
* Presence of one or more of the following conditions: type 2 diabetes or hypertension. (Type 2 diabetes and hypertension will be defined by the combination of a self-reported physician diagnosis of one of the conditions and at least one pharmacy prescription for one of the conditions.)
* Able to converse, and complete the research surveys in English or Spanish, based on self-report.
* Positive screening for food or nutrition insecurity by:

  1. Hunger Vital Sign™ screening and,
  2. Nutrition Security Screener

Exclusion Criteria:

* Unable to provide informed consent.
* Unable to read and write.
* Self-reported serious medical conditions that may be expected to shorten life expectancy to less than one year
* A condition that limits participant's ability to grocery shop or choose food for themselves
* Plans to move to a new home in the next 6 months that would require use of a different pharmacy
* Currently pregnant or pregnancy planned within the next 6 months
* Currently using or planning to start an insulin pump or other automated insulin delivery device within the next 6 months
* Currently on a GLP-1 agonist or planning to start a GLP-1 agonist within the next 6 months
* Currently receiving or planning to receive within the next 6 months another Food is Medicine program, like PRx, Grocery Rx, or Medically Tailored Meals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of PRx Program Utilization | Up to 6-months
  The utilization rate will be calculated by dividing the number of PRx cards redeemed by the total number of PRx cards distributed at each pharmacy.
Rate of PRx Program Redemption | Up to 6-months
  The redemption rates will be calculated based on the average proportion of dollar amounts redeemed over the total dollar amounts of benefits distributed.
Change in Food Security | baseline, 3-months, 6-months
  Assessed by the USDA's Household Food Security Survey Module: Six-Item Short Form. The sum of affirmative responses to the six questions is the household's raw score. A raw score of 0-1 indicates food security, while a score of 2-6 indicates food insecurity.
Change in Nutrition Security | baseline, 3-months, 6-months
  Assessed by the Nutrition Security Screener. Respondents will be classified as nutrition secure if they answer, "Not hard at all" or "Not very hard" to item 1 or nutrition insecure if they answer, "Somewhat hard", "Hard", or "Very Hard."
Change in Diet Quality | baseline, 3-months, 6-months
  Assessed by a modified Mini-Eating Assessment Tool (EAT). A calculated score will be created such that a higher score is indicative of healthier dietary patterns.

SECONDARY OUTCOMES:
Change in Hemoglobin A1c | baseline and 6-months
  For participants with diabetes, pharmacy staff will conduct a point-of-care hemoglobin A1c measurement of blood obtained by fingerstick.
Change in Continuous Glucose Monitor (CGM) Time-in-range | baseline and 6-months
  Time-in-range is the percentage of time spent with glucose levels in the target range. For participants with diabetes, pharmacy staff place a CGM, per product instructions, on the participant with a goal to wear for 10 days (each time).
Change in Blood Pressure | baseline and 6-months
  Pharmacy staff will measure participants' systolic and diastolic blood pressure.
Change in Body Mass Index | baseline and 6-months
  Pharmacy staff will collect height and weight.
Change in Patient Reported Health Related Quality of Life | baseline, 3-months, 6-months
  Assessed by PROMIS (Patient-Reported Outcomes Measurement Information System) Global Health, the scoring system converts responses from a 10-item questionnaire into T-scores for Global Physical Health (GPH) and Global Mental Health (GMH), where higher scores indicate better health.
Change in Disease Self-management | baseline, 3-months, 6-months
  Assessed by the 6-item Self Efficacy for Managing Chronic Disease (SEMCD) scale. Scores will be calculated as the mean response to the six questions. A higher score is indicative of higher self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Dariush Mozaffarian, MD, DrPH, Principal Investigator — The Food is Medicine Institute at the Friedman School of Nutrition Science and Policy at Tufts University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Information Website — https://tuftsfoodismedicine.org/project/nacds/
- See also: Eligibility Website — https://sites.tufts.edu/cp3study/